CLINICAL TRIAL: NCT01812915
Title: Comparison of Tapered- vs. Cylindrical-shaped Tube Cuffs Pressure Alteration With Nitrous Oxide Diffusion Under General Anesthesia
Brief Title: Comparison of Tapered- vs. Cylindrical-shaped Tube Cuffs Pressure Alteration With Nitrous Oxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Junyong In, MD, Associate Professor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: J In 2013-1
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Adverse Effect of Other General Anesthetics; Anesthesia Intubation Complication; Inhalation of Nitrous Oxide; Trachea
Keywords: Cuff pressure; Cylindrical cuff; Endotracheal tube; Nitrous oxide; Tapered cuff
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cylindrical-shape cuff ETT (Group C) (Experimental): Control group: Mallinckrodt HiLo(TM) endotracheal tube. Intracuff pressures of the tubes every 10 minutes, Adult patients under general anesthesia with Mallinckrodt Hi-Lo(TM) tube.
  Interventions: Device: Cylindrical-shape cuff ETT (Group C)
- Tapered-shape cuff ETT (Group T) (Experimental): Experimental group: Mallinckrodt TaperGuard(TM) endotracheal tube. Intracuff pressures of the tubes every 10 minutes, Adult patients under general anesthesia with Mallinckrodt TaperGuard(TM) tube.
  Interventions: Device: Tapered-shape cuff ETT (Group T)

INTERVENTIONS:
Device: Cylindrical-shape cuff ETT (Group C) — Randomized allocation of the endotracheal cuffs for general anesthesia, mechanical ventilation will be maintained with Mallinckrodt Hi-Lo(TM) endotracheal tube.
  Other Names: Mallinckrodt Hi-Lo(TM) endotracheal tube
  Arms: Cylindrical-shape cuff ETT (Group C)
Device: Tapered-shape cuff ETT (Group T) — Randomized allocation of the endotracheal cuffs for general anesthesia, mechanical ventilation will be maintained with Mallinckrodt TaperGuard(TM) endotracheal tube.
  Other Names: Mallinckrodt TaperGuard(TM) endotracheal tube
  Arms: Tapered-shape cuff ETT (Group T)

SUMMARY:
When using nitrous oxide for general anesthesia, nitrous oxide diffusion induces intracuff hyperinflation of the endotracheal tube. Furthermore the difference among various types of cuffed endotracheal tubes in cuff pressure behavior during nitrous oxide exposure.

TaperGuard(TM) tube has been newly introduced and has tapered-shape cuff. In vitro study, the intracuff pressure of TaperGuard(TM) tube was lower than that of conventional tube with cylindrical-shaped cuff of the conventional tube(Hi-Lo(TM) tube). Therefore, this clinical study is needed to evaluate the intracuff pressure during general anesthesia with nitrous oxide exposure.

DETAILED DESCRIPTION:
During 60 minutes after routine anesthetic induction and intubation of the endotracheal tubes, intracuff pressures will be measured every 10 minutes with a manometer (VBM, Sulz, Germany).

60% nitrous oxide will be added at time 0. For 60 minutes from the beginning of general anesthesia, intracuff pressures will be measured every 10 minutes.

After 60 minutes, Intracuff pressures will be maintained around 20 cm H2O during the remaining period of the surgery.

The questionnaire for a sore throat, hoarseness, and dysphagia will be questioned at about 1, 6, and 24 hours after the surgery and the general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo general anesthesia in a supine position with a neutral position of the head (hand and forearm sugery)
* 18~70 years old
* American society of anesthesiologists physical status 1-2
* Body mass index < 30 kg/m2

Exclusion Criteria:

* Contraindication for nitrous oxide
* Difficult intubation
* Cormack-Lehane grade > 3
* Airway-related or pulmonary diseases
* Short or long operation time (< 1 hour or > 3 hours)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Intracuff pressure of the endotracheal tube after 60 min (1 hour) with exposure to nitrous oxide | One hour after the exposure to nitrous oxide under general anesthesia

SECONDARY OUTCOMES:
Intracuff pressure of the endotracheal tubes | 0, 10, 20, 30, 40, 50 minutes after exposure to nitrous oxide
  Intracuff pressures will be measured with a manometer (VBM, Sulz, Germany)
Postoperative sore throat: incidence | About 1, 6, 24 hours after termination of anesthesia
Postoperative hoarseness: incidence | About 1, 6, 24 hours after termination of anesthesia
Postoperative dysphagia: incidence | About 1, 6, 24 hours after termination of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Junyong In, M.D., Ph.D., Principal Investigator — DongGuk University
Locations (1):
- Dongguk University Ilsan Hospital, Goyang, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsuboi S, Miyashita T, Yamaguchi Y, Yamamoto Y, Sakamaki K, Goto T. The TaperGuard endotracheal tube intracuff pressure increase is less than that of the Hi-Lo tube during nitrous oxide exposure: a model trachea study. Anesth Analg. 2013 Mar;116(3):609-12. doi: 10.1213/ANE.0b013e318279b399. Epub 2013 Feb 11. PMID 23400983